CLINICAL TRIAL: NCT06606158
Title: Rehabilitation in Total Hip Arthroplasty Through a Mobile Application: A Retrospective Observational Study
Brief Title: Rehabilitation in Total Hip Arthroplasty Through a Mobile Application
Acronym: HIP-App
Status: Completed | Type: Observational
Sponsor: Universidad Pontificia Comillas (Other)
Responsible Party: Principal Investigator, Joaquín Zambrano Martín, MSc, Universidad Pontificia Comillas
Other Study IDs: UPC-EIDUM24/25
Record Dates: First submitted 2024-07-15; First posted 2024-09-20 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Total Hip Arthroplasty
Keywords: Hip Prosthesis; Mobile Applications; Rehabilitation Programs; Digital Health; Patient Reported Outcome Measures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Non-exposed cohort (mobile application follow-up considered as a protective factor).: Patients who, following hip arthroplasty surgery, were monitored using a mobile application designed to record physical activity data and adherence to a postoperative recovery exercise program. Patients received scheduled instructions regularly within the application, providing educational material and exercise/activity routines, but did not receive formal physical therapy outside of the application as part of the study.
  Interventions: Other: App exercises program
- Cohort 2: Exposed cohort (no mobile application follow-up).: Patients who, following hip arthroplasty surgery, did not undergo follow-up via the mobile application and followed the standard recovery protocol, which includes regular clinic visits and conventional physiotherapy.
  Interventions: Other: Exercises program

INTERVENTIONS:
Other: Exercises program — Strength, mobility, and balance exercises described within the standardized Physiotherapy plan.
  Groups: Cohort 2: Exposed cohort (no mobile application follow-up).
Other: App exercises program — A strength, mobility, and balance exercise program delivered through a mobile app.
  Groups: Cohort 1: Non-exposed cohort (mobile application follow-up considered as a protective factor).

SUMMARY:
This observational retrospective study aims to assess the rehabilitation outcomes of patients who underwent total hip arthroplasty (THA) and were monitored through a mobile application versus those who were not. The hypothesis is that patients who receive postoperative follow-up via a mobile app, which includes a recovery exercise program, will experience significantly greater improvements in functionality, quality of life, and treatment adherence compared to those who do not use the app after three months of follow-up.

The study will analyze the records of patients from two cohorts: one group monitored with the mobile application and another group receiving standard postoperative care without the app. Data on patients' functionality, quality of life, and adherence to treatment will be collected and compared between the two groups. This study seeks to provide evidence on the effectiveness of digital health interventions in enhancing postoperative recovery for THA patients.

DETAILED DESCRIPTION:
This study adopts an observational, analytical, longitudinal, and retrospective design with two cohorts: an exposed cohort and a non-exposed cohort, aimed at evaluating the effectiveness of a follow-up program using a mobile application in patients undergoing total hip arthroplasty.

Patients selected for this study have undergone total hip arthroplasty using the Furlong Evolution® short stem and acetabular cup prosthetic design (ACE). Surgeries were performed at Hospital San Juan de Dios de Santurtzi and Hospital Universitario de Galdakao, both located in Vizcaya.

To analyze the new care model (functional recovery program and patient follow-up via a digital application), the entire study population from June 1, 2023, to March 30, 2024, will be included, conducting a complete cohort analysis with a 3-month follow-up period.

Data collection includes sociodemographic, clinical, and pre-surgical functional characteristics. Specific assessment tests were employed to evaluate pain, function, and quality of life.

Electronic health records will be used to collect data, including demographic variables (age, gender), medical history, Patient-Reported Outcome Measures (PROMs) such as the Harris Hip Score and WOMAC scale and Patient-Reported-Experience-Mesures (PREMs) as satisfaction scale.

Quality assurance procedures will be implemented to ensure data validity and registry integrity, including data validation checks, source data verification against external sources, and a comprehensive data dictionary detailing each variable's origin and coding information.

Standard Operating Procedures (SOPs) will guide registry operations, including patient recruitment, data collection, management, analysis, adverse event reporting, and change management.

A statistical analysis plan will employ appropriate analytical principles and techniques to address primary and secondary objectives outlined in the study protocol, assessing the sample size required to demonstrate significant effects and strategies for handling missing data.

This detailed description encompasses the comprehensive framework and methodology of the study, emphasizing rigorous data collection, quality assurance measures, and statistical analysis strategies essential for evaluating the effectiveness of the mobile application-based follow-up program in post-total hip arthroplasty patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old operated at Hospital San Juan de Dios de Santurtzi and Hospital Universitario de Galdakao, both located in Vizcaya.
* Operated on for total hip arthroplasty with the Furlong Evolution short stem prosthetic design and ACE acetabular cup.
* Patients who have started postoperative rehabilitation program with or without the mobile application.
* Ability to walk before the fracture with or without the aid of instruments or persons.
* Access to a smartphone with the ability to install applications.
* Patients with complete PROMs data using the Harris Hip Score and WOMAC scale available.

Exclusion Criteria:

* Patients with incomplete data or lack of follow-up at three months.
* Patients with severe comorbidities that may significantly affect mobility and functionality.
* Patients with cognitive impairment that precludes the use of the mobile application for recovery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing total hip arthroplasty: Patients were selected who underwent total hip arthroplasty using the same prosthetic design, Furlong Evolution® short stem and ACE acetabular cup. Surgeries were performed at Hospital San Juan de Dios de Santurtzi and Hospital Universitario de Galdakao, both located in Vizcaya.
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Harris Hip Score (HHS) | Evaluation using the HHS is conducted preoperatively, and subsequently at 1 month and 3 months following hip arthroplasty surgery for each participant.
  The HHS is a widely used metric to evaluate functional status and hip-related quality of life in patients undergoing total hip arthroplasty. It measures functional capacity based on pain, gait, mobility, and ability to perform daily activities.
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Assessment using the WOMAC Index occurs pre-hip arthroplasty surgery, and again at 1 and 3 months post-surgery for each study participant.
  The WOMAC Index is a validated measure assessing pain, stiffness, and physical function in hip osteoarthritis patients. It provides a detailed evaluation of functional disability and impact on hip-related quality of life.

SECONDARY OUTCOMES:
Satisfaction Scale | Assessment using a visual analog scale at 1 and 3 months post-surgery for each participant in the study.
  A visual analog scale is used in which the patient simultaneously evaluates their degree of pain and satisfaction, in addition to providing their perception of health status, functional capacity, changes in pain intensity, the impact of arthroplasty on their well-being, and whether their expectations of the surgery have been met

CONTACTS AND LOCATIONS:
Overall Officials: Joaquín Zambrano-Martín, MSc, Principal Investigator — International School of Doctoral Studies, University of Murcia, Murcia, Spain; Comillas Pontifical University, Health Sciences, Department. San Juan de Dios School of Nursing and Physical Therapy, Madrid, Spain
Locations (1):
- International School of Doctoral Studies, University of Murcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No